CLINICAL TRIAL: NCT00651742
Title: An Open-Label, Non-Randomized, Multicenter, Two-Stage, Phase 2 Study of S-1 in Chemotherapy-Naïve Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Phase 2 Study of S-1 in Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry); United BioSource, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1204
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- S-1 30 mg/m^2 (Experimental): Participants received 30 milligrams per meter square (mg/m^2) of S-1 orally twice daily (BID) for 2 weeks (i.e., Day 1 to 14), followed by 1 week recovery period (i.e., Day 15 to 21; one cycle equaled 21 days), treatment was repeated every 3 weeks until death, progression of disease, occurrence of intolerable side effects, withdrawal of consent, or removal by Investigator, whichever comes first.
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — All participants received S-1 orally at a dose of 30 mg/m2 BID for 14 days followed by a 1-week recovery period, repeated every 3 weeks. The trial was planned to proceed to the second stage only if sufficient efficacy was demonstrated in Stage 1.

SUMMARY:
The purpose of this study is to determine whether S-1 is effective in slowing tumor activity in participants with locally advanced or metastatic pancreatic cancer who have not had chemotherapy. The study is also looking at the safety of S-1.

DETAILED DESCRIPTION:
Locally advanced or metastatic pancreatic cancer is relatively unresponsive to chemotherapy. This is true for the nucleoside analogue gemcitabine, with a response rate of approximately 10%, as well as for 5-fluorouracil (5-FU). Even when gemcitabine is combined with other chemotherapeutic drugs or biological agents, the overall tumor response rate remains basically unchanged. S-1 is a new generation oral fluoropyrimidine that combines Tegafur (5-fluoro-1-(tetrahydro-2-furanyl)-2,4(1H,3H)-pyrimidinedione [FT]), an oral prodrug of 5-FU, with two modulators, Gimeracil (5-chloro-2,4-dihydroxypyridine [CDHP]), which inhibits 5-FU degradation by dihydropyrimidine dehydrogenase (DPD) inhibition, and Oteracil potassium (Oxo), which inhibits 5-FU phosphorylation in the digestive tract. This combination of 3 compounds is designed to achieve enhanced antitumor activity while decreasing gastrointestinal toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent.
2. Has histologically or cytologically confirmed locally advanced, unresectable or metastatic adenocarcinoma of the pancreas not amenable to curative radiotherapy or surgery.
3. Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (ie, lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20 mm using conventional techniques or ≥ 10 mm using spiral computed tomography [CT] scan).
4. Is able to take medications orally.
5. Is 18 years of age or older.
6. Has a Karnofsky Performance Status (KPS) ≥ 70%.
7. Has a life expectancy of ≥ 12 weeks.
8. Has adequate organ function as defined by the following criteria:

   1. Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times the upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastasis, then AST (SGOT) and ALT (SGPT) may be ≤ 5 times ULN.
   2. Total serum bilirubin ≤ 3.0 times ULN (if due to underlying liver metastasis, then total bilirubin may be ≤ 5 times ULN).
   3. Absolute granulocyte count ≥ 1,500/mm3 (ie, ≥ 1.5 x 109/L by International Units [IU]).
   4. Platelet count ≥ 100,000/mm3 (IU: ≥ 100 x 109/L).
   5. Hemoglobin value ≥ 9.0 g/dL.
   6. Calculated creatinine clearance ≥ 60 mL/min (based on serum creatinine) (Cockcroft-Gault85 formula)
9. Is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Has had treatment with any of the following within the specified time frame prior to study drug administration:

   1. Any prior anticancer chemotherapy.
   2. Radiation therapy to a target lesion unless there was evidence of PD after radiotherapy (and this target lesion must not be the only site of measurable disease).
   3. Any radiotherapy within the previous 3 weeks.
   4. Any investigational agent received either concurrently or within the last 30 days.
   5. Current enrollment in another clinical study with an investigational agent. Patients participating in surveys or observational studies are eligible to participate in this study.
2. Major surgery within the previous 3 weeks.
3. Symptomatic brain metastasis not controlled by corticosteroids.
4. Leptomeningeal metastasis.
5. Previous or concurrent malignancy other than pancreatic cancer except adequately treated carcinoma in-situ of the cervix or non-melanoma skin cancer.
6. Uncontrolled ascites requiring drainage at least twice a week.
7. Other serious illness or medical condition(s) including, but not limited to, the following:

   1. Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class III or IV), angina pectoris, arrhythmias, or hypertension.
   2. Active infection.
   3. Known (at time of entry) gastrointestinal disorder, including malabsorption, chronic nausea, vomiting, or diarrhea, present to the extent that it might interfere with oral intake and absorption of study medication.
   4. Poorly controlled diabetes mellitus.
   5. Psychiatric disorder that may interfere with consent and/or protocol compliance.
   6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
   7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
8. Is receiving a concomitant treatment with drugs interacting with S-1. The following drugs are prohibited because there may be an interaction with S-1:

   1. Sorivudine, uracil, cimetidine, folinic acid, and dipyridamole (may enhance S-1 activity).
   2. Allopurinol (may diminish S-1 activity).
   3. Phenytoin (S-1 may enhance phenytoin activity).
   4. Flucytosine, a fluorinated pyrimidine antifungal agent (may enhance S-1 and flucytosine activity).
9. Is a pregnant or lactating female.
10. Has known sensitivity to 5-FU.
11. Is a patient with reproductive potential who refuses to use an adequate means of contraception (including male patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-01-09 (Actual); Primary Completion 2008-07-08 (Actual); Study Completion 2008-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Central, Study Director — Taiho Oncology, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 centers in the Germany between 09-January-2006 to 08-July-2008.
Pre-assignment Details: The enrollment of Stage 2 of the study was not initiated, as sufficient efficacy per protocol was not demonstrated in Stage 1. Overall, 29 participants were screened, of them 28 participants were enrolled and 27 received study treatment in Stage 1.
Period: Overall Study
Arm/Group | S-1 30 mg/m^2
Started (Enrolled) | 28
Treated | 27
Efficacy Analysis Per Investigator | 21
Efficacy Analysis Per Independent Reader | 25
Completed | 0
Not Completed | 28
Not completed — Objective Disease Progression | 22
Not completed — Toxicity | 3
Not completed — Investigator Judgment | 1
Not completed — Withdrawal of Consent | 1
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received at least one dose of study treatment.
Groups:
- S-1 30 mg/m^2: Participants received 30 mg/m^2 of S-1 orally BID for 2 weeks (i.e., Day 1 to 14), followed by 1 week recovery period (i.e., Day 15 to 21; one cycle equaled 21 days), treatment was repeated every 3 weeks until death, progression of disease, occurrence of intolerable side effects, withdrawal of consent, or removal by Investigator, whichever comes first.
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response Rate (ORR)
Description: ORR was defined as the percentage of participants with objective evidence of partial response (PR) or complete response (CR) and was based on the best overall response across all cycles for each participant. Tumor response was assessed according to the Response Evaluation Criteria In Solid Tumors (RECIST). For target lesions response, CR was defined as the disappearance of all target lesions for at least 3 weeks and PR was defined as at least a 30% reduction in the sum of the longest diameters of the target lesions, taking as a reference the baseline sum of the longest diameters for at least 6 weeks. For non-target lesions, CR was defined the disappearance of all non-target lesions and normalization of tumor marker level for at least 6 weeks.
Time Frame: From first dose of study medication until disease progression, permanent discontinuation of study treatment, or death due to any cause, assessed up to 2 years 5 months
Population: Primary efficacy population included all participants in the safety population who met the key eligibility criteria (1st line therapy in participants with measurable pancreatic locally advanced or metastatic disease) and had at least one response assessment after starting study treatment. Here, 'Number analyzed' signifies number of participants in the specified population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
percentage of participants
  Independent Assessment: number analyzed (Participants) | 25
  Independent Assessment | 4.0 [0.1 to 20.4]
  Investigator Assessment: number analyzed (Participants) | 21
  Investigator Assessment | 9.5 [1.2 to 30.4]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with objective evidence of CR, PR or stable disease (SD) determined according to RECIST. For target lesions, stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as a reference the smallest sum of the longest diameters since the treatment started for at least 6 weeks. For non-target lesions, stable disease was defined a persistence of greater than or equal to (>=) 1 non-target lesions and/or maintenance of tumor marker level above the normal limits for at least 6 weeks.
Time Frame: as for outcome 1
Population: Analysis was performed on primary efficacy population. Here, 'Number analyzed' signifies number of participants in the specified population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
percentage of participants
  Independent Assessment: number analyzed (Participants) | 25
  Independent Assessment | 68.0 [46.5 to 85.1]
  Investigator Assessment: number analyzed (Participants) | 21
  Investigator Assessment | 76.2 [52.8 to 91.8]

3. Secondary Outcome: Duration of Response (DR)
Description: DR was calculated as date of first progressive disease (PD) or death, date after the first response of CR or PR minus date of first CR or PR plus 1. Participants who did not die and were without progressive disease were censored at last evaluable tumor response assessment. Analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Analysis was performed on primary efficacy population. Here, 'Number analyzed' signifies number of participants evaluable in specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
months
  Independent Assessment: number analyzed (Participants) | 25
  Independent Assessment | 7.4 [NA to NA] — Upper and lower limit of Confidence Interval (CI) is not estimable, due to less number of participants with event.
  Investigator Assessment: number analyzed (Participants) | 21
  Investigator Assessment | NA [2.8 to NA] — Median and upper limit of CI is not estimable, due to less number of participants with event.

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was calculated as date of first PD minus date of first dose of study medication plus 1. Participants without progressive disease were censored at last evaluable tumor response assessment. Analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Analysis was performed on primary efficacy population. Here, 'Number analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
months
  Independent Assessment: number analyzed (Participants) | 25
  Independent Assessment | 3.5 [1.6 to 5.5]
  Investigator Assessment: number analyzed (Participants) | 21
  Investigator Assessment | 3.5 [2.5 to 5.3]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated as date of death minus date of first dose of study medication plus 1. In the absence of death confirmation, OS was censored at the date of last study follow-up. Analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Analysis was performed on safety population that included all the participants who had received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
months | 9.1 [4.7 to 11.2]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as date of first PD or date of death minus date of first dose of study medication plus 1. Participants who did not die and were without PD were censored at their last evaluable tumor response assessment. Analysis was performed by Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
months
  Independent Assessment: number analyzed (Participants) | 25
  Independent Assessment | 3.5 [1.6 to 5.5]
  Investigator Assessment: number analyzed (Participants) | 21
  Investigator Assessment | 3.5 [2.5 to 5.3]

7. Secondary Outcome: Number of Participants With Karnofsky Performance Status (KPS) Score - Shift From Baseline Score to Final Assessment Score
Description: KPS classified participant's as per their functional impairment. The KPS ranged from 0percent (%) to 100%, (100= no signs of disease, 90% = few symptoms or signs of disease, 80%=some symptoms or signs, 70% = not capable of normal activity or work, 60% = can take care of most personal requirements, 50% = requires frequent medical care, 40% = disabled, 30% = severely disabled, hospital admission indicated but no risk of death, 20% = very ill, requires supportive measures or treatment, 10% = moribund, rapidly progressive fatal disease processes, and 0% = death), where higher values represented better outcomes. Participants with baseline KPS >=70% were included in study. Final assessment was the participant's last assessment. Participants with available data were only presented in the below data table.
Time Frame: Baseline, at end of treatment (up to 2 years 5 months)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
Participants
  Baseline score 100% shift to Final assessment score 100% | 6
  Baseline score 100% shift to Final assessment score 90% | 7
  Baseline score 100% shift to Final assessment score 70% | 1
  Baseline score 100% shift to Final assessment score 0% | 1
  Baseline score 90% shift to Final assessment score 90% | 1
  Baseline score 90% shift to Final assessment score 80% | 3
  Baseline score 90% shift to Final assessment score 70% | 1
  Baseline score 90% shift to Final assessment score 60% | 1
  Baseline score 90% shift to Final assessment score 0% | 2
  Baseline score 80% shift to Final assessment score 80% | 1
  Baseline score 80% shift to Final assessment score 0% | 2
  Baseline score 70% shift to Final assessment score 0% | 1

8. Secondary Outcome: Change From Baseline in Pain Intensity
Description: Pain intensity was graded from 0 (least possible pain) to 100 (worst possible pain) on a visual analog scale (VAS). The higher score on VAS scale indicated more pain. Final assessment was the last assessment of participant's.
Time Frame: Baseline, at end of treatment (up to 2 years 5 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
millimeters (mm) | -6.47 (27.619)

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical event in a participants administered any dose of a study medication which may or may not have a causal relationship with the use of the study medication. An SAE was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event.
Time Frame: From the first dose of study medication up to 30 days after the last dose of study medication, or until additional antitumor therapy had been introduced, whichever came first (approximately up to 2 years 6 months)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | S-1 30 mg/m^2
Number analyzed (Participants) | 27
Participants
  At Least 1 AE | 25
  At Least 1 SAE | 15

ADVERSE EVENTS:
Time Frame: From the first dose of study medication up to 30 days after the last dose of study medication, or until additional antitumor therapy had been introduced, whichever came first (approximately up to 2 years 6 months).
Description: Analysis was performed on safety population that included all the participants who had received at least one dose of study medication.
Arm/Group | S-1 30 mg/m^2
All-Cause Mortality (participants affected / at risk) | 24/27
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1 30 mg/m^2 (N=27)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 4 (4)
Fatigue (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1 30 mg/m^2 (N=27)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 4 (6)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 2 (3)
Conjunctivitis (Eye disorders) | 3 (3)
Lacrimation increased (Eye disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Ascites (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 10 (15)
Pancreatic insufficiency (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 9 (13)
Asthenia (General disorders) | 2 (2)
Chills (General disorders) | 3 (3)
Fatigue (General disorders) | 10 (13)
General physical health deterioration (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (6)
Hepatic pain (Hepatobiliary disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3)
Blood creatinine increased (Investigations) | 2 (2)
Blood urea increased (Investigations) | 3 (4)
Haemoglobin decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 9 (9)
Weight increased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6)
Vitamin k deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Since the pre-defined tumor response futility criteria was not exceeded in Stage 1, participant enrollment for Stage 2 was not conducted, as pre-planned in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes